CLINICAL TRIAL: NCT03405519
Title: MR-guided RAdiotherapy to Breast With Dose Escalation to regionaL Lymph NodEs
Acronym: MIRABELLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR4738
Record Dates: First submitted 2018-01-10; First posted 2018-01-23 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy planning (Other): Radiotherapy planning using both CT and MRI scans
  Interventions: Procedure: Radiotherapy planning using both CT and MRI scans

INTERVENTIONS:
Procedure: Radiotherapy planning using both CT and MRI scans — Patients' radiotherapy will be planned using CT and MRI scans in order to establish the best methodology for planning of radiotherapy for nodal disease

SUMMARY:
Radiotherapy to the breast and lymph nodes is routinely planned using CT scans. The introduction of magnetic resonance imaging (MRI) has the potential to better visualise the lymph nodes and so define a smaller treatment area or 'target'. This means that the dose delivered to the target could be increased without increasing the dose to normal tissues. The MIRABELLE study is designed to test if this is possible by recruiting patients diagnosed with breast cancer including lymph node disease. The investigators will ask participants to have a CT scan and an MRI scan before they have radiotherapy. The investigators will then plan radiotherapy using both these scans and compare the possible dose delivered to the lymph nodes using the MRI and CT defined lymph nodes. This will not affect the patient's future treatment.

DETAILED DESCRIPTION:
MR imaging has the potential to improve both the localisation of pan-LN treatments and the subsequent treatment delivery using MR-linac technology. The MIRABELLE study will apply the MR sequences developed in LN-negative volunteers/patients to the context of node-positive breast cancer patients with the aim of reducing the delineated nodal volume thereby facilitating dose-escalation to involved LNs. The benefit of using MRI for LN localisation as compared to conventional CT imaging will be investigated by determining whether a higher dose can be delivered using MRI- as compared to CT-based delineation. Any increase in dose will be deemed a success as this has potential to improve tumour control. In addition, inter-observer errors in outlining will be explored to investigate whether these are reduced using MRI. Reduced inter-observer errors would result in smaller margins for error such that less normal tissue could be irradiated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Female or male
* Invasive carcinoma of the breast (left or right-sided)
* cT1-T4,N3,M0-1 disease
* Due to proceed to primary treatment (chemo, surgery, radiotherapy and/or endocrine therapy)
* Histopathological involvement of axillary lymph nodes confirmed on FNA or Bx
* Likely to undergo locoregional radiotherapy as part of their breast cancer management

Exclusion Criteria:

* Implanted pacemakers and/or pacing wires
* Cochlear implants
* Programmable hydrocephalus shunts
* Implanted neurostimulation systems
* Implanted drug infusion pumps
* Ferromagnetic implants
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
The number of patients in whom a higher dose can be delivered to the level IV (SCF) nodes without breaching brachial plexus constraints on the radiotherapy plans created using MR images compared with CT images | During a radiotherapy planning process, an average of 2 weeks
  MR images are acquired with patient in a position as close as possible to the radiotherapy CT planning position. Images are acquired in a radiotherapy CT scanner with patient in a position replicating that achieved in the MRI scanner. The images are imported into a treatment planning system and consensus lymph node volume agreed between an expert radiation oncologist and MR radiologist. All pan-LN will be delineated on co-registered MRI sequences and on CT (using ESTRO guidelines) by 7 observers.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kirby, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided